CLINICAL TRIAL: NCT00457860
Title: A Phase 1, Multicenter, Dose Escalation Study of CAT-8015 in Patients With Relapse or Refractory Chronic Lymphocytic Leukemia (CLL), Prolymphocytic Leukemia (PLL), or Small Lymphocytic Lymphoma (SLL)
Brief Title: Safety Study of CAT-8015 Immunotoxin in Patients With CLL, PLL or SLL With Advance Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge Antibody Technology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1002; NCT00453284 (obsolete NCT alias)
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Leukemia
Keywords: CLL; PLL; SLL; Relapse; Refractory; immunotoxin; HA22; CAT-8015; immunotherapy
MeSH Terms: conditions — Leukemia; Recurrence | interventions — immunotoxin HA22; Biological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Immunotoxin therapy
Drug: CAT-8015 immunotoxin
Procedure: Biological therapy

SUMMARY:
RATIONALE: The CAT-8015 immunotoxin can bind tumor cells and kill them without harming normal cells. This may be an effective treatment for chronic lymphocytic leukemia (CLL), prolymphocytic leukemia (PLL), or small lymphocytic lymphoma (SLL that has not responded to chemotherapy, surgery or radiation therapy.

PURPOSE: Phase I dose escalation study to determine the maximum tolerated dose of CAT-8015 immunotoxin in treating patients who have chronic lymphocytic leukemia, prolymphocytic leukemia or small lymphocytic lymphoma that has not responded to treatment

DETAILED DESCRIPTION:
OUTLINE: Patients receive CAT-8015 IV over 30 minutes on days 1, 3, and 5 followed by rest. Treatment repeats every 4 weeks for up to a total of 10 courses in the absence of dose limiting toxicity, complete response or disease progression. Patients are followed at 1, 3, 6,12,15,18, 21, 24 months following the start of the last treatment cycle.

Cohorts of 3-6 patients each will receive escalating doses of recombinant CAT-8015 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose proceeding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, between16 to 25 new patients will be added to the MTD cohort depending on how well the CAT-8015 is tolerated.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell leukemia (CLL, PLL or SLL)
* Measurable disease
* Patients with chronic lymphocytic leukemia (CLL), or small lymphocytic lymphoma (SLL) are eligible if they have failed 2 or more prior courses of standard chemotherapy and/or biologic therapy (e.g. Rituxan) and if treatment for progressive disease is medically indicated. Patients with prolymphocytic leukemia (PLL) will be eligible if they have failed at least one prior standard chemotherapeutic regimen. Medical indications for treatment include progressive disease-related symptoms, progressive cytopenias due to marrow involvement, progressive or painful splenomegaly or adenopathy, rapidly increasing lymphocytosis, autoimmune hemolytic anemia or thrombocytopenia and increased frequency of infections.

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Life expectancy of greater than 6 months, as assessed by the principal investigator

Other

* Patients with other cancers who meet eligibility criteria and have had less than 5 years of disease-free survival will be considered on a case-by-case basis
* Ability to understand and sign informed consent
* Female and male patients agree to use an approved method of contraception during the study

EXCLUSION CRITERIA:

* Documented and ongoing central nervous system involvement with their malignant disease (history of CNS involvement is not an exclusion criterion)
* History of bone marrow transplant
* Pregnant or breast-feeding females
* Patients whose plasma contains either a significant level of antibody to CAT-8015 as measured by ELISA, or antibody that neutralizes the binding of CAT-8015 to CD22 as measured by a competition ELISA.
* HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs)
* Hepatitis B surface antigen positive
* Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements

Hepatic function: serum transaminases (either ALT or AST) or direct bilirubin:

* ≥ Grade 2, unless bilirun is due to Gilbert's disease

Renal function: serum creatinine clearance ≤60mL/min as estimated by Cockroft-Gault formula

Hematologic function:

* The ANC <1000/cmm, or platelet count <50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy)
* Baseline coagulopathy > grade 3 unless due to anticoagulant therapy
* A patient will not be excluded because of pancytopenia ≥ Grade 3, or erythropoietin dependence, if it is due to disease, based on the results of bone marrow studies

Pulmonary function:

* Patients with < 50% of predicted forced expiratory volume (FEV1) or <50% of predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin concentration and alveolar volume. Note: Patients with no prior history of pulmonary illness are not required to have PFTs. FEV1 will be assessed following bronchodilator therapy.

Recent prior therapy:

* Cytotoxic chemotherapy, corticosteriods (except stable doses of prednisone), whole body electron beam radiation therapy, hormonal, biologic or other systemic therapy or investigational therapy of the malignancy for 3 weeks prior to entry into the trial
* Less than or equal to < 3 months prior monoclonal antibody therapy (i.e. rituximab)
* Patients who have received or are receiving radiation therapy less than 3 weeks prior to study entry will be not be excluded providing the volume of bone marrow treated is less than 10% and also the patient has measurable disease outside the radiation port

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2007-03

PRIMARY OUTCOMES:
Estimate the maximum dose that can be safely administered to a patient
Characterize the toxicity profile of CAT-8015
Study the clinical pharmacology of CAT-8015
Observe anti-tumor activity, if any

SECONDARY OUTCOMES:
To assess the potential of CAT-8015 to induce antibodies
To Investigate the potential of biomarkers to predict any therapeutic or toxic response

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Warren Grant Megnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
- Klinika Hemtologii Uniwersytetu Medycznego (Medical University of Lodz), Lodz, Poland

REFERENCES:
- [Background] Kreitman RJ, Squires DR, Stetler-Stevenson M, Noel P, FitzGerald DJ, Wilson WH, Pastan I. Phase I trial of recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) in patients with B-cell malignancies. J Clin Oncol. 2005 Sep 20;23(27):6719-29. doi: 10.1200/JCO.2005.11.437. Epub 2005 Aug 1. PMID 16061911